CLINICAL TRIAL: NCT00523497
Title: Noninvasive Mechanical Ventilation in Severe Community-Acquired Pneumonia and Acute Hypoxemic Respiratory Failure. A Prospective, Randomized and Controlled Study
Brief Title: Efects of Noninvasive Mechanical Ventilation and Conventional Mechanical Ventilation in Patients With Severe Comunity Pneumonia
Acronym: NIMV AND SCAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis of the present study showed a significant decrease in mortality rate (p= 0.04) as well as in the number of days at the ICU p=0.0002.
Sponsor: Hospital Privado del Sur (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NIV67-07
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Last update posted 2007-08-31 (Estimated); Status verified 2007-08

CONDITIONS: Community Acquired Pneumonia.; Acute Hypoxemic Respiratory Failure
Keywords: Severe community-acquired pneumonia; Noninvasive mechanical ventilation; Acute hypoxemic respiratory failure.
MeSH Terms: conditions — Community-Acquired Pneumonia; Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Non invasive mechanical ventilation

SUMMARY:
The purpose of this study is to determine whether the noninvasive ventilation is more effective in the treatment of severe comunity acquired pneumonia in comparison with the conventional mechanical ventilation with orotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

The criteria for the diagnosis of SCAP included:

* Blood systolic pressure lower than 90 mmHg or blood diastolic pressure lower than 60 mmHg
* RR higher than 30 breaths per minute
* PaO2/FiO2 lower than 250 while breathing through a Venturi mask with a 50% inspired oxygen fraction (FiO2)
* Bilateral or multiple lobar infiltrations evidenced by thorax X-ray, and
* Use of vasopressor drugs

Exclusion Criteria:

Exclusion criteria included:

* COPD
* Asthma
* Acute cardiogenic pulmonary edema
* Severe haemodynamic instability (arterial systolic pressure lower than 70 mmHg) or requirements of vasoactive drugs
* Glasgow score equal to or lower than 9 or requiring OTI for airway protection or for recent pulmonary resucitation
* Antecedents of respiratory failure resulting from neuromuscular pathology
* Failure of two or more organs
* Facial deformities; and
* Recent facial, aesophagic and gastric surgeries

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
The primary aim of this study was to compare the effects of NIMV on mortality rate and length of stay at the ICU with the effects of CMV | 3 years

SECONDARY OUTCOMES:
The secondary aims were to evaluate the incidence and the complications of OTI as well as to compare the improvements in the gas exchange. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: S. A Lasdica, Study Principal Investigator, Principal Investigator
Locations (1):
- Hospital Privado del Sur, Bahía Blanca, Buenos Aires, Argentina